CLINICAL TRIAL: NCT05870579
Title: A Phase Ib Dose Finding Study Assessing Safety and Activity of [177Lu]Lu-NeoB in Combination With Ribociclib and Fulvestrant in Participants With Estrogen Receptor Positive, Human Epidermal Growth Factor Receptor-2 Negative and Gastrin Releasing Peptide Receptor Positive Advanced Breast Cancer Experiencing Early Relapse From (Neo)Adjuvant Endocrine Therapy or Who Have Progressed on Endocrine Therapy in Combination With a CDK4/6 Inhibitor for Advanced Disease
Brief Title: [177Lu]Lu-NeoB in Combination With Ribociclib and Fulvestrant in Participants With ER+, HER2- and GRPR+ Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAA603B12101; 2022-502465-18-00 (Other: EU CTIS)
Record Dates: First submitted 2023-05-08; First posted 2023-05-23 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Advanced breast cancer; Radioligand therapy; Ribociclib; Fulvestrant; Lutetium; NeoB; Estrogen receptor (ER); ER-positive; Human epidermal growth factor 2 (HER2); HER-2 negative; Gastrin releasing peptide receptor (GRPR); GRPR-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Fulvestrant; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Participants will receive [177Lu]Lu- NeoB in combination with ribociclib and fulvestrant, in the dose escalation and the backfill parts of the study. Goserelin administration is only applicable for pre/peri-menopausal women and men.
  Interventions: Drug: [68Ga]Ga-NeoB; Drug: [177Lu]Lu-NeoB; Drug: Ribociclib; Drug: Fulvestrant; Other: Goserelin

INTERVENTIONS:
Drug: [68Ga]Ga-NeoB — [68Ga]Ga-NeoB serves as a radioactive imaging compound to be used for PET imaging for localization of GRPR positive lesions, at screening, potentially at Cycle 2 Day 15 visit, and between 4 and 8 weeks after the last administered dose of [177Lu]Lu-NeoB.
  [68Ga]Ga-NeoB will be administered as a single intravenous (i.v.) dose.
  Other Names: gallium neoB
Drug: [177Lu]Lu-NeoB — Study participants will receive [177Lu]Lu-NeoB once every cycle
  Other Names: lutetium neoB
Drug: Ribociclib — 600 mg once daily (OD) days 1 to 21 every 28 days
  Other Names: kisqali
Drug: Fulvestrant — 500 mg at Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and every 28 days thereafter
Other: Goserelin — For pre/peri-menopausal women and men only.
  Other Names: zoladex

SUMMARY:
The purpose of this trial is to estimate the recommended dose (RD) of [177Lu]Lu-NeoB in combination with ribociclib and fulvestrant in participants with estrogen receptor (ER) positive (ER+), human epidermal growth factor receptor-2 (HER2) negative (HER2-) and gastrin releasing peptide receptor (GRPR) positive (GRPR+) advanced breast cancer experiencing early relapse from (neo)adjuvant endocrine therapy or who have progressed on endocrine therapy in combination with a CDK4/6 inhibitor for advanced disease.

DETAILED DESCRIPTION:
The study comprises of a dose escalation part and, a concurrent backfill part.

1. The dose escalation part will estimate the RD of [177Lu]Lu-NeoB in combination with ribociclib and fulvestrant; four provisional dose levels are planned to be tested: 100 millicurie (mCi) (initial dose), 150mCi, 200 mCi and 250mCi in cohorts of 3 to 6 participants. After inclusion of each cohort of 3 to 6 participants, the incidence rate of DLTs will be compared to the pre-defined toxicity rate boundaries to decide whether the next cohort will receive a lower, higher or same dose or whether the trial will be terminated.
2. The backfill part will allow enrollment to a previously cleared dose level (during escalation part) in order to obtain additional safety, tolerability as well as preliminary efficacy data. During the backfill part, the cumulative incidence rate of DLTs will also be compared to the pre-defined toxicity rate boundaries to determine if escalation should be restarted from a lower dose level.
3. The recommended dose (RD) will be determined considering all available data from the escalation and backfill part.

During screening, study participants will receive the investigational imaging agent [68Ga]Ga-NeoB. An additional administration of the [68Ga]Ga-NeoB will be performed potentially at Cycle 2 Day 15, and within 4-8 weeks from the last administration of [177Lu]Lu-NeoB for a positron emission tomography (PET)/computed tomography (CT) or PET/magnetic resonance imaging (MRI). Study treatment will include [177Lu]Lu-NeoB on day 1 of each 28-day cycle (+ =< 3 days) for 6 cycles, ribociclib (once daily; days 1 to 21 in a 28-day cycle) and fulvestrant (C1D1, C1D15, C2D1 and every 28 days thereafter) until disease progression. Pre- and perimenopausal women and men will additionally receive goserelin on day 1 of every cycle.

During the treatment period participants will be required to attend a site visit approximately every 28 days, on the first day of each cycle (as well as on C1D2, C1D3, C1D8, C1D15, C2D15, C3D3 and C5D3), to undergo study treatment administration, dosimetry and safety assessments. Tumor assessments are performed every 8 weeks until month 18, every 12 weeks until month 36 and as clinically indicated thereafter, until disease progression. After study treatment discontinuation, participants will be followed up for safety for 8 weeks after their last study treatment administration. Beyond the initial 8 weeks of safety follow-up, all participants will be followed up every 12 weeks until month 36 and every 24 weeks thereafter until month 60 for a total of 5 years from the participant's enrollment in the study, or until death, lost to follow-up, or withdrawal of consent (WoC), whichever occurs first.

The end of study is defined as the date of the last visit, scheduled procedure or follow up (or date of death, WoC or lost to follow up, whichever occurs first) of the last participant in the study globally, or at 5 years from the date of the last participant enrolled, whichever occurs earlier.

ELIGIBILITY:
Key Inclusion criteria:

* Adult female or male >= 18 years of age at the time of informed consent
* Histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive with ER >10% (regardless of progesterone receptor (PgR) expression) breast cancer by local laboratory testing (based on the most recently analyzed tissue sample)
* HER2 negative breast cancer defined as a negative in situ hybridization test or an immunohistochemistry (IHC) status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (e.g. fluorescence in situ hybridization (FISH), chromogenic in situ hybridization (CISH), or silver in situ hybridization (SISH)) test is required by local laboratory testing (based on the most recently analyzed tissue sample)
* Participant has advanced (loco regionally recurrent not amenable to curative therapy (e.g. surgery and/or radiotherapy) or metastatic) breast cancer

Participants may be:

1. relapsed with documented evidence of relapse on or within 12 months from completion of (neo)adjuvant endocrine therapy (+/- CDK4/6 inhibitor) with no treatment for advanced disease OR
2. relapsed with documented evidence of relapse more than 12 months from completion of (neo)adjuvant endocrine therapy and then subsequently progressed with documented evidence of progression after one line of endocrine therapy (except fulvestrant) (+/- CDK4/6 inhibitor) for advanced disease OR
3. advanced breast cancer at diagnosis that progressed with documented evidence of progression after one line of endocrine therapy (except fulvestrant) (+/- CDK4/6 inhibitor) Note: Participant who relapsed with documented evidence of relapse on/or within 12 months from completion of (neo)adjuvant endocrine therapy and then subsequently progressed with documented evidence of progression after one line of endocrine therapy (with either an antiestrogen or an aromatase inhibitor) for advanced disease will NOT be included in the study. At least one target lesion (i.e., a measurable lesion as per RECIST 1.1) in the baseline stand-alone CT or MRI, showing [68Ga]Ga-NeoB uptake on PET/CT or PET/MRI scoring 2 or higher, based on the Visual Scoring Scale.

   * Adequate bone marrow and organ function as defined by the laboratory values.
   * Standard 12-lead ECG values defined as the mean of the triplicate ECGs and assessed locally:
   * QT interval corrected by Fridericia's formula (QTcF) interval at screening < 450 msec
   * Mean resting heart rate 50-90 bpm (determined from the ECG)
   * Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Key Exclusion criteria:

* More than one line of prior treatment in the advanced/metastatic setting. Participant shouldn't have received prior fulvestrant treatment.
* Documented evidence of prior ribociclib dose reduction due to safety reasons either in adjuvant setting or for advanced disease.
* Relapse or disease progression within 6 months of receiving a CDK4/6 inhibitor therapy either in adjuvant setting or for advanced disease. Symptomatic visceral disease or any disease burden that makes the participant ineligible for ribociclib plus endocrine treatment per the Investigator's best judgment.
* Presence of central nervous system (CNS) involvement unless meeting BOTH of the following criteria: 1) At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment. 2) Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme inducing anti-epileptic medications for brain metastases.
* Currently receiving warfarin or other Coumadin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin, or fondaparinux is allowed.
* Diagnosis of inflammatory breast cancer at screening
* Child Pugh score B or C
* History or current diagnosis of impaired cardiac function, clinically significant cardiac disease or ECG abnormalities indicating significant risk of safety for participants.
* Known or expected hypersensitivity to any of the study drugs or any of their excipients.
* Prior administration of a radiopharmaceutical unless 10 or more half-lives have elapsed before injection of [68Ga]Ga-NeoB or [177Lu]Lu-NeoB
* Participant has received extended-field RT=< 4 weeks or limited field RT=< 2 weeks prior to start of treatment and has not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia or other toxicities not considered a safety risk for the participant at Investigator's discretion) and/or prior external beam radiation therapy (EBRT) to more than 25% of the bone marrow.
* Participant is currently receiving or has received systemic corticosteroids =< 2 weeks prior to starting study treatment, or who have not fully recovered from side effects of such treatment. Note: The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
* Participant has a history of or ongoing acute pancreatitis within 1 year of screening.
* Participant is currently receiving any of the following substances and cannot be discontinued 7 days prior to starting study treatment:
* Concomitant medications, herbal supplements, and/or fruits (e.g., grapefruit, pummelos, star fruit, Seville oranges) and their juices that are strong inducers or inhibitors of cytochrome P450 (CYP) 3A4
* Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
* Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointes (TdP) that cannot be discontinued or replaced by safe alternative medication (e.g., within 5 half-lives or 7 days prior to starting study treatment)
* Participant is currently receiving NEP inhibitors (e.g.Entresto®, racecadotril) and images for dosimetry assessments cannot be acquired for this participant.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2032-01-26 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of DLTs during the DLT observation period | 28 days after the first administration of [177Lu]Lu-NeoB
  A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness/injury, or concomitant medications that occurs within the DLT period from C1D1 of treatment with [177Lu]Lu-NeoB, ribociclib and fulvestrant with or without goserelin. The National Cancer Institute (NCI) CTCAE version 5.0 will be used for all grading.
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | From date of enrollment till 8 weeks after end of Treatment, assessed up to approximately 60 months
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Incidence of dose interruptions, discontinuation and dose reductions | From date of enrollment till 8 weeks after end of Treatment, assessed up to approximately 60 months
  Dose interruptions, discontinuation and dose reductions will be assessed for tolerability.

SECONDARY OUTCOMES:
Time activity curves (TACs) of [177Lu]Lu-NeoB in organs and tumor lesions | Cycles 1, 3 and 5: Day 1 (1-4 hours post-dose/post-infusion (p.i.)), Day 2 (24 hours p.i), Day 3 (48 hours p.i), Day 8 (168 hours p.i) (1 cycle = 4 weeks)
  Time activity curves (TACs) for the various organs and lesions will be produced as percentage of injected dose in selected organs and lesions.
Absorbed radiation doses of [177Lu]Lu-NeoB in organs and tumor lesions | Cycles 1, 3 and 5: Day 1 (1-4 hours post-dose/post-infusion (p.i.)), Day 2 (24 hours p.i), Day 3 (48 hours p.i), Day 8 (168 hours p.i) (1 cycle = 4 weeks)
  The absorbed dose in target organs will be summarized with descriptive statistics.
Concentration of [177Lu]Lu-NeoB in blood over time | Cycle 1: Day 1 (Pre-dose (before start of infusion), At end of infusion, 0.5, 1, 2, 4 and 6 hours post-dose/post-infusion (p.i.)), Day 2 (24 hours p.i), Day 3 (48 hours p.i), Day 8 (168 hours p.i)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. Blood concentration of [177Lu]Lu-NeoB will be summarized with descriptive statistics.
Observed maximum blood concentration (Cmax) of [177Lu]Lu-NeoB | Cycle 1: Day 1 (Pre-dose (before start of infusion), At end of infusion, 0.5, 1, 2, 4 and 6 hours post-dose/post-infusion (p.i.)), Day 2 (24 hours p.i), Day 3 (48 hours p.i), Day 8 (168 hours p.i)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. Cmax will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) of [177Lu]Lu-NeoB | Cycle 1: Day 1 (Pre-dose (before start of infusion), At end of infusion, 0.5, 1, 2, 4 and 6 hours post-dose/post-infusion (p.i.)), Day 2 (24 hours p.i), Day 3 (48 hours p.i), Day 8 (168 hours p.i)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. Tmax will be listed and summarized using descriptive statistics.
Area under the blood concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of [177Lu]Lu-NeoB | Cycle 1: Day 1 (Pre-dose (before start of infusion), At end of infusion, 0.5, 1, 2, 4 and 6 hours post-dose/post-infusion (p.i.)), Day 2 (24 hours p.i), Day 3 (48 hours p.i), Day 8 (168 hours p.i)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. AUClast will be listed and summarized using descriptive statistics.
Total systemic clearance for intravenous administration (CL) of [177Lu]Lu-NeoB | Cycle 1: Day 1 (Pre-dose (before start of infusion), At end of infusion, 0.5, 1, 2, 4 and 6 hours post-dose/post-infusion (p.i.)), Day 2 (24 hours p.i), Day 3 (48 hours p.i), Day 8 (168 hours p.i)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. CL will be listed and summarized using descriptive statistics.
Volume of distribution during the terminal phase following intravenous elimination (Vz) of [177Lu]Lu-NeoB | Cycle 1: Day 1 (Pre-dose (before start of infusion), At end of infusion, 0.5, 1, 2, 4 and 6 hours post-dose/post-infusion (p.i.)), Day 2 (24 hours p.i), Day 3 (48 hours p.i), Day 8 (168 hours p.i)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. Vz will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T^1/2) of [177Lu]Lu-NeoB | Cycle 1: Day 1 (Pre-dose (before start of infusion), At end of infusion, 0.5, 1, 2, 4 and 6 hours post-dose/post-infusion (p.i.)), Day 2 (24 hours p.i), Day 3 (48 hours p.i), Day 8 (168 hours p.i)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. T^1/2 will be listed and summarized using descriptive statistics.
Objective Response Rate (ORR) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 60 months
  Objective Response Rate (ORR) is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR), as per local review and according to RECIST 1.1.
Duration of Response (DoR) | From first documented evidence of CR or PR (the response prior to confirmation) until time of documented disease progression or death due to any cause, whichever comes first, assessed up to approximately 60 months
  Duration of Response (DOR) was defined as the duration between the date of first documented Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) and the date of first documented radiographic progression or death due to any cause as per local review and according to RECIST 1.1.
Time to Response (TTR) | From the date of first dose to the date of documented response (CR or PR), assessed up to approximately 60 months
  Time to response (TTR) is the time from the date of first dose of [177Lu]Lu-NeoB to the first documented response (CR or PR) according to RECIST 1.1.
Clinical Benefit Rate (CBR) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 60 months
  Clinical Benefit Rate (CBR) is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) or maintaining an overall response of Stable Disease (SD) for at least 24 weeks. CR, PR, and SD are defined as per local review according to RECIST 1.1.
Progression Free Survival (PFS) | From the date of first dose to the date of confirmed progression or death due to any cause, whichever comes first, assessed up to approximately 60 months
  Progression Free Survival (PFS) is defined as the time from the date of first dose of [177Lu]Lu-NeoB to the date of confirmed progression or death due to any cause. PFS will be assessed via local review according to RECIST 1.1.
Overall Survival (OS) | From the date of first dose to date due to any cause, assessed up to approximately 60 months
  Overall Survival (OS) is defined as the time from date of first dose of [177Lu]Lu-NeoB to date of death due to any cause.
Incidence and severity of AEs following [68Ga]Ga-NeoB administration | 3 days after [68Ga]Ga-NeoB administration
  Incidence and severity of AEs following [68Ga]Ga-NeoB administration at screening will be done via the analysis of frequencies for Adverse Event (AEs), Serious Adverse Event (SAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- United States (6):
  - UCLA Jonsson Comp Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of Kansas Medical Center, Westwood, Kansas
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Utah Intermountain Medical Center, Murray, Utah
- China (3):
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- France (5):
  - Novartis Investigative Site, Saint-Cloud, Hauts De Seine
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
- Germany (4):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
- Novartis Investigative Site, Gliwice, Poland
- Novartis Investigative Site, Porto, Portugal
- Spain (4):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taunk NK, Escorcia FE, Lewis JS, Bodei L. Radiopharmaceuticals for Cancer Diagnosis and Therapy: New Targets, New Therapies-Alpha-Emitters, Novel Targets. Cancer J. 2024 May-Jun 01;30(3):218-223. doi: 10.1097/PPO.0000000000000720. PMID 38753757